CLINICAL TRIAL: NCT05637905
Title: The Predictive Value of Monocyte Chemoattractant Protein -1 in the Development of Cardiovacular Events in Psoriatic Arthritis Patients
Brief Title: Monocyte Chemoattractant Protein-1 in Psoriatic Arthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Anas Mostafa Mohamed, doctor, Assiut University
Other Study IDs: MCP-1
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psoriatic arthritis patients group
- health control group

SUMMARY:
1. Evaluate serum levels of (MCP-1) in PsA with or without cardiovascular affaction .
2. Detect subclinical cardiovascular affaction in patients with PsA for early diagnosis and management .

DETAILED DESCRIPTION:
Psoriatic arthritis (PSA) is an autoimmune disease arising from the interply between proinflamatory cytokines

[1]and external stimuli in genetically predisposed individuals.[2]

* The disease is chronic and affects the peripheral joints and may include axial skeleton with or without extrarticular manifestations.[3]
* Abnormal activation of the innate and adaptive immune systems contributes to chronic disease processes in both psoriasis and PSA .[4] The skin and the joints exhibit a prominent lymphocytic infiltrate consisting of activated CD4+ and CD8+ T cells as well as an increase in neutrophil infiltration[5].

Patients with PsA have a higher risk of developing a cardiovascular(CV) events than the general population. This could be attributed to the higher prevalence of traditional cardiovascular risk factors and to the disease characteristics such as systemic inflammation. [6] These patients may show asymptomatic cardiomyopathy even in the absence of traditional risk factors [7].Cardiac dysfunction is associated with a poor prognosis, increased mortality, and affact socioecenomic function of patients therefore, the diagnosis of the cardiac dysfunction in the asymptomatic phase of the disease [8] is important for the timely introduction of therapy [9].Monocyte chemotactic protien1(MCP-1) is a member of chemotactic chemokines(CC) which are secreted by immune effector cells and dysfunctional endothelium [10].

* The pivotal function of MCP-1 is to attract monocyte in the arterial wall through increased expression of adhesion molecules on their surface that interacts with endothelium[11].
* MCP-1 induce maturation of monocyte in the arterial wall ,which then become specialized macrophage in early atheroma and produce tissue factors supporting coagulation and proinflammatory cytokines such as IL-1 and IL-6. It affects the functions of the surrounding immune effector cells in locally thickened intima.[12]
* During active disease in psoriatic skin lesions and synovial tissue, activated monocytes represent the major source of proinflammatory mediators, including the chemokine MCP-1 [13]. MCP-1 is thought to be involved in the pathogenesis of oedema and bone erosion in patients with PsA [14].

ELIGIBILITY:
Inclusion Criteria:

* PsA patients (age ≥ 18years) who fulfilled the CASPAR classification criteria[15]for psoriatic arthritis

Exclusion Criteria:

* PsA patients with

  1. infection.
  2. bone marrow disorders.
  3. other autoimmune diseases.
  4. diabetes.
  5. hypertention .
  6. hyperlipidemia.
  7. liver diseases.
  8. renal diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: psoriatic arthritis patients with or without clinically cardiovascular affaction
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
MCP-1 | two month
  :Evaluate serum levels of monocyte chemoattractant protein-1(MCP-1) in relation to echocardiographic changes in patient with psoriatic arthritis.

SECONDARY OUTCOMES:
Echocardiography | two month
  b.Detect subclinical cardiovascular affaction in patient with psoriatic arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Abass, doctor, Study Director — Assiut University; Mohamed Raouf, doctor, Study Director — Assiut University; Esraa Ahmed, doctor, Study Director — Assiut University

REFERENCES:
- See also: 1.V.Chandran,F.Abji,A.V. Perruccio et al.,"Serum-basedsoluble markers difffferentiate psoriatic arthritis from osteoarthritis," Annals of the Rheumatic Diseases,vol.78, no.6, pp.796-801,2019. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: A. L. Carvalho and C. M. Hedrich, "The molecular pathophysiology of psoriatic arthritis-the complex interplay between genetic predisposition, epigenetics factors, and the microbiome," Frontiers in Molecular Biosciences, vol. 8, p. 662047, 2021. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: A. B. Gottlieb and J. F. Merola, "Axial psoriatic arthritis: an update for dermatologists," Journal of the American Academy of Dermatology, vol. 84, no. 1, pp. 92-101, 2021 — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: Lories RJ, de Vlam K. Is psoriatic arthritis a result of abnormalities in acquired or innate immunity? Curr Rheumatol Rep 2012; 14: 375-382. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: .Lowes MA, Kikuchi T, Fuentes-Duculan J, Cardinale I, Zaba LC, Haider AS, et al. Psoriasis vulgaris lesions contain discrete populations of Th1 and Th17 T cells. J Invest Dermatol 2008; 128: 1207-12 — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: Risk Reclassification According to Cardiovascular Six Traditional Cardiovascular Risk Algorithms and a Carotid Ultrasound in Psoriatic Arthritis Patients — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: A. Rana, V. K. Mahajan, K. S. Mehta et al., "Cardiomyopathy and echocardiographic abnormalities in Indian patients with psoriasis: results of a pilot study," International Journal of Clinical Practice, vol. 75, no. 3, p. e13756, 2021. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: P. S. Pagel, J. N. Tawil, B. T. Boettcher et al., "Heart failure with preserved ejection fraction: a comprehensive review and update of diagnosis,pathophysiology, treatment, and perioperative implications," Journal of Cardiothoracic and Vascular Anesthes — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: .E. L. Potter, S. Ramkumar, H. Kawakami et al., "Association of asymptomatic diastolic dysfunction assessed by left atrial strain with incident heart failure,"JACC: Cardiovascular Imaging, vol. 13, no. 11, pp. 2316-2326, 2020. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: Lin, V. Kakkar, and X. Lu, "Impact of MCP -1 in atherosclerosis," Current Pharmaceutical Design, vol. 20, no. 28, pp. 4580-4588, 2014. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: C. Papadopoulou, V. Corrigall, P. R. Taylor, and R. N. Poston, "The role of the chemokines MCP-1, GRO-α, IL-8 and their receptors in the adhesion of monocytic cells to human atherosclerotic plaques," Cytokine, vol. 43, no. 2, pp. 181-186, 2008. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: P. Aukrust, B. Halvorsen, A. Yndestad et al., "Chemokines and cardiovascular risk," Arteriosclerosis, Thrombosis, and Vascular Biology, vol. 28, no. 11, pp. 1909-1919 — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: D. E. Furst and J. S. Louie, "Targeting inflammatory pathways in axial spondyloarthritis," Arthritis Research & Therapy, vol. 21, no. 1, p. 135, 2019. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: Y. R. Woo, C. J. Park, H. Kang, and J. E. Kim, "The risk of systemic diseases in those with psoriasis and psoriatic arthritis:from mechanisms to clinic," International Journal of Molecular Sciences, vol. 21, no. 19, p. 7041, 2020. — http://pubmed.ncbi.nlm.nih.gov/30910989/
- See also: .Moll JM, Wright V Psoriatic arthritis. Semin Arthritis Rheum 1973;3:55-78.CrossRefPubMedGoogle Scholar. — http://pubmed.ncbi.nlm.nih.gov/30910989/